CLINICAL TRIAL: NCT02452528
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Multi-dose Study to Determine the Depth of Hepatitis B Surface Antigen (HBsAg) Reduction Following Intravenous ARC-520 in Combination With Entecavir or Tenofovir in Patients With HBeAg Positive, Chronic Hepatitis B Virus (HBV) Infection
Brief Title: Study of ARC-520 in Participants With Hepatitis B Virus e Antigen (HBeAg) Positive Chronic Hepatitis B Virus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Company decision to discontinue trial
Sponsor: Arrowhead Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Heparc-2004
Record Dates: First submitted 2015-05-15; First posted 2015-05-22 (Estimated); Results first posted 2017-11-01 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Chronic Hepatitis B
Keywords: Hepatitis B Virus; Chronic Hepatitis B; HBV
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B | interventions — ARC-520; entecavir; Tenofovir; Diphenhydramine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ARC-520 (Experimental): Intravenous administration of 1.0 mg/kg ARC-520 once every 4 weeks for 3 total doses, plus entecavir (0.5 or 1.0 mg/day) or tenofovir (300 mg/day), taken throughout the study.
  Pretreatment with diphenhydramine 50 mg 2 hours (±30 minutes) prior to administration of study drug.
  Interventions: Drug: ARC-520; Drug: Entecavir; Drug: Tenofovir; Drug: diphenhydramine
- Placebo (Placebo Comparator): Intravenous administration of normal saline (0.9%) once every 4 weeks for 3 total doses, plus entecavir (0.5 or 1.0 mg/day) or tenofovir (300 mg/day), taken throughout the study.
  Pretreatment with diphenhydramine 50 mg 2 hours (±30 minutes) prior to administration of placebo.
  Interventions: Drug: Placebo; Drug: Entecavir; Drug: Tenofovir; Drug: diphenhydramine

INTERVENTIONS:
Drug: ARC-520
  Arms: ARC-520
Drug: Placebo
  Arms: Placebo
Drug: Entecavir — 0.5 or 1.0 mg/day orally
  Other Names: Baraclude
Drug: Tenofovir — 300 mg/day orally
  Other Names: Viread
Drug: diphenhydramine — 50 mg orally as pretreatment antihistamine

SUMMARY:
Participants with chronic HBV infection will receive multiple doses of ARC-520 in combination with entecavir or tenofovir and be evaluated for safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 to 75 years of age
* Written informed consent
* Body mass index (BMI) between 17.5 and 30.0 kg/m2
* No clinically significant abnormalities at screening/pre-dose 12-lead ECG assessment
* No abnormal finding of clinical relevance
* Diagnosis of HBeAg positive, immune active, chronic HBV infection
* > 2 months of continuous treatment with daily oral entecavir or tenofovir
* Must use 2 effective methods of contraception (double barrier contraception or hormonal contraceptive along with a barrier contraceptive)

Exclusion Criteria:

* Pregnant or lactating
* Acute signs of hepatitis/other infection within 4 weeks of screening
* Hepatic transaminases (alanine aminotransferase [ALT] or aspartate aminotransferase [AST]) > 3 times the upper limits of normal
* Liver Elastography (i.e. FibroScan®) score > 9
* Antiviral therapy other than entecavir or tenofovir within 3 months of screening
* Prior treatment with interferon in the last 3 years
* Use of anticoagulants, corticosteroids, immunomodulators, or immunosuppressants within 6 months of screening
* Use within 7 days prior to screening of dietary and/or herbal supplements that can interfere with liver metabolism
* Use of any drugs known to induce or inhibit hepatic drug metabolism within 30 days of study drug administration
* Use of prescription medication within 14 days prior to study drug administration
* Depot injection/implant of any drug except birth control within 3 months prior to study drug administration
* Known diagnosis of diabetes mellitus
* History of autoimmune disease
* Human immunodeficiency virus (HIV) infection
* Sero-positive for Hepatitis C Virus (HCV), and/or a history of delta virus hepatitis
* Hypertension; blood pressure > 150/100 mmHg
* History of cardiac rhythm disturbances
* Family history of congenital long QT syndrome, Brugada syndrome or unexplained sudden cardiac death
* Symptomatic heart failure, unstable angina, myocardial infarction, severe cardiovascular disease within 6 months prior to study entry
* History of malignancy, except for adequately treated basal cell carcinoma, squamous cell skin cancer, superficial bladder tumors, in situ cervical cancer
* Major surgery within 3 months of screening
* History of alcohol and/or drug abuse < 12 months from screening
* Regular use of alcohol within 6 months (ie, more than 14 units of alcohol per week)
* Evidence of systemic acute inflammation, sepsis, or hemolysis
* Diagnosed with a significant psychiatric disorder
* Use of drugs of abuse
* History of allergy to bee venom
* Positive reaction to the bee venom allergy immunoglobulin E (IgE) test
* Use of investigational agents or devices within 30 days
* Clinically significant inherited or acquired gastrointestinal pathology, unresolved gastrointestinal symptoms, liver or kidney disease
* Presence of cholangitis, cholecystitis, cholestasis, or duct obstruction
* Clinically significant history or presence of uncontrolled systemic disease
* Donated or had a loss of whole blood of 50 milliliters (mL) to 499 mL within 30 days or more than 499 mL between 31 and 56 days prior to study treatment
* History of fever within 2 weeks of screening
* Immunization/planned immunization with live attenuated vaccine except influenza vaccine
* Presence of any medical or psychiatric condition or social situation that impacts compliance or results in additional safety risk
* Excessive exercise/physical activity within 7 days of screening/enrolment or during study
* History of coagulopathy/stroke within past 6 months, and/or concurrent anticoagulant medication(s)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-08; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Research Site 1, San Francisco, California
  - Research Site 2, Miami, Florida
  - Research Site 4, New York, New York
  - Research Site 6, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ARC-520 | Placebo
Started | 2 | 2
Completed | 1 | 1
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ARC-520 | Placebo | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 0 | 1 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Quantitative Hepatitis B Surface Antigen (Log qHBsAg) at Day 85
Time Frame: Baseline, Day 85
Population: At the time of study termination only 2 ARC-520-treated and 2 placebo-treated participants had been enrolled. Due to the small sample size, analysis of this primary endpoint was not performed.
Arm/Group | ARC-520 | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), Deaths, and Discontinuations Due to Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a participant which does not necessarily have to have a causal relationship with treatment. An SAE was defined as any untoward medical occurrence that, at any dose: results in death; is life-threatening; requires inpatient hospitalization or prolongation of an existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; or is a medically important event or reaction. An AE was classified as a TEAE if the AE was not present prior to the first study medication administration and started at or after the time of initiation of administration of study medication, or if the AE presented prior to initiation of administration of study medication, continued and increased in intensity after administration of study medication.
Time Frame: From time of informed consent through Day 147 ± 3 days
Population: All participants who received at least 1 dose of ARC-520 or placebo
Measure: Count of Participants; unit: Participants
Arm/Group | ARC-520 | Placebo
Number analyzed (Participants) | 2 | 2
Participants
  TEAEs | 0 | 1
  SAEs | 0 | 0
  Deaths | 0 | 0
  Discontinuations due to AEs | 0 | 0

3. Secondary Outcome: Pharmacokinetics of ARC-520: Area Under the Plasma Concentration-Time Curve From Time 0 to 24 Hours (AUC0-24)
Time Frame: Through 48 hours post-dosing on Days 1 and 57
Population: Pharmacokinetic evaluation was to be performed only on participants receiving ARC-520. At the time of study termination only 2 ARC-520-treated participants had been enrolled and therefore pharmacokinetic samples were not processed and no statistical analysis was performed.
Arm/Group | ARC-520 | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Pharmacokinetics of ARC-520: Area Under the Plasma Concentration-Time Curve From Time 0 to the Last Quantifiable Plasma Concentration (AUClast)
Time Frame: Through 48 hours post-dosing on Days 1 and 57
Population: as for outcome 3
Arm/Group | ARC-520 | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Pharmacokinetics of ARC-520: Area Under the Plasma Concentration-Time Curve From Time 0 Extrapolated to Infinity (AUCinf)
Time Frame: Through 48 hours post-dosing on Days 1 and 57
Population: Pharmacokinetic evaluation was to be performed only on participants receiving ARC-520. At the time of study termination only 2 ARC-520 treated participants had been enrolled and therefore pharmacokinetic samples were not processed and no statistical analysis was performed.
Arm/Group | ARC-520 | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Pharmacokinetics of ARC-520: Maximum Observed Plasma Concentration (Cmax)
Time Frame: Through 48 hours post-dosing on Days 1 and 57
Population: as for outcome 5
Arm/Group | ARC-520 | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Pharmacokinetics of ARC-520: Apparent Clearance (CL)
Time Frame: Through 48 hours post-dosing on Days 1 and 57
Population: as for outcome 5
Arm/Group | ARC-520 | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Pharmacokinetics of ARC-520: Apparent Volume of Distribution (V)
Time Frame: Through 48 hours post-dosing on Days 1 and 57
Population: as for outcome 5
Arm/Group | ARC-520 | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Pharmacokinetics of ARC-520: Terminal Elimination Rate Constant (Kel)
Time Frame: Through 48 hours post-dosing on Days 1 and 57
Population: as for outcome 5
Arm/Group | ARC-520 | Placebo
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Pharmacokinetics of ARC-520: Terminal Elimination Half-Life (t1/2)
Time Frame: Through 48 hours post-dosing on Days 1 and 57
Population: as for outcome 5
Arm/Group | ARC-520 | Placebo
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Pharmacokinetics of Entecavir or Tenofovir: AUC0-24
Time Frame: Through 24 hours post-dosing on Days 1 and 57
Population: as for outcome 5
Arm/Group | ARC-520 | Placebo
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Pharmacokinetics of Entecavir or Tenofovir: AUClast
Time Frame: Through 24 hours post-dosing on Days 1 and 57
Population: as for outcome 5
Arm/Group | ARC-520 | Placebo
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Pharmacokinetics of Entecavir or Tenofovir: Cmax
Time Frame: Through 24 hours post-dosing on Days 1 and 57
Population: Pharmacokinetic evaluation was to be performed only on subjects receiving ARC-520. At the time of study termination only 2 ARC-520 treated subjects had been enrolled and therefore pharmacokinetic samples were not processed and no statistical analysis was performed.
Arm/Group | ARC-520 | Placebo
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Pharmacokinetics of Entecavir or Tenofovir: Time of Cmax (Tmax)
Time Frame: Through 24 hours post-dosing on Days 1 and 57
Population: as for outcome 5
Arm/Group | ARC-520 | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From time of informed consent through Day 147 ± 3 days
Arm/Group | ARC-520 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 1/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARC-520 (N=2) | Placebo (N=2)
Fatigue (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No